CLINICAL TRIAL: NCT00004088
Title: Sequential High-Dose Melphalan and Busulfan/Cyclophosphamide Followed by Peripheral Blood Progenitor Cell Rescue, Interferon/Thalidomide and Pamidronate for Patients With Multiple Myeloma
Brief Title: Combination Chemo, Peripheral Stem Cell Transplant, Biological Therapy, Pamidronate and Thalidomide for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99021; P30CA033572 (NIH); CHNMC-IRB-99021 (Other: City of Hope Institutional Review Board); NCI-G99-1583 (Other: National Cancer Institute); CDR0000067301 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2018-01

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Interferon-alpha; Introns; Busulfan; Cyclophosphamide; Melphalan; Pamidronate; Thalidomide; Peripheral Blood Stem Cell Transplantation

ARMS (1):
- HD chemotherapy followed by PBPC Rescue (Experimental): Patients receive high-dose (HD) melphalan intra-venously (IV) on day -1. Peripheral blood progenitor cells (PBPCs) are reinfused on day 0. Filgrastim (G-CSF) is administered IV or SC daily beginning on day 1 and continuing until blood counts recover. Between 8 and 14 weeks later, patients receive IV high-dose busulfan every 6 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2. PBPCs are reinfused on day 0 and G-CSF is administered IV or subcutaneously (SC) daily until blood counts recover.
  Interventions: Biological: filgrastim; Biological: recombinant interferon alfa; Drug: busulfan; Drug: cyclophosphamide; Drug: melphalan; Drug: pamidronate disodium; Drug: thalidomide; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
  Other Names: granulocyte colony-stimulating factor (G-CSF); Neupogen
Biological: recombinant interferon alfa
  Other Names: IFN alpha-2B; Intron A
Drug: busulfan
  Other Names: Myleran; Busulfex
Drug: cyclophosphamide
  Other Names: cytophosphane; Cytoxan
Drug: melphalan
  Other Names: Alkeran; Evomela
Drug: pamidronate disodium
  Other Names: pamidronic acid
Drug: thalidomide
  Other Names: Thalidomid; Immunoprin
Procedure: peripheral blood stem cell transplantation
  Other Names: peripheral blood progenitor cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy drugs and kill more cancer cells. Biological therapies, such as interferon alfa, use different ways to stimulate the immune system and stop cancer cells from growing. Thalidomide may stop the growth of cancer cells by stopping blood flow to the tumor. Pamidronate may help to reduce the side effects of treatment for multiple myeloma.

PURPOSE: This phase II trial is studying combination chemotherapy, peripheral stem cell transplantation, biological therapy, pamidronate, and thalidomide to see how well they work in treating patients with stage I, stage II, or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and toxic effects of high-dose melphalan, busulfan, and cyclophosphamide followed by autologous peripheral blood stem cell rescue, interferon alfa, and pamidronate in patients with responsive or stable, low-bulk multiple myeloma.
* Determine the response rate and progression-free and overall survival of patients treated with this regimen.
* Determine the feasibility of adding thalidomide to interferon alfa and pamidronate in patients who are not in complete remission (CR) 6 months after the second course of high-dose chemotherapy.
* Determine whether administration of thalidomide can increase the CR rate in patients who are not in CR 6 months after the second course of high-dose chemotherapy and determine its effect on progression-free and overall survival of these patients.
* Determine the pharmacokinetics of busulfan and cyclophosphamide and correlate the pharmacokinetics with the toxic effects of these drugs and outcome in these patients.
* Determine the effect of thalidomide on microvascular density of bone marrow and correlate these possible effects with outcome in these patients.
* Determine the cytogenetics, gene rearrangement, and fluorescence in situ hybridization in baseline and post treatment bone marrow and blood specimens and correlate the presence/persistence of these features with treatment outcome in these patients.

OUTLINE: Patients receive cyclophosphamide IV over 2 hours on day 1 and filgrastim (G-CSF) subcutaneously (SC) or IV twice a day beginning on day 2 and continuing until peripheral blood stem cells (PBSCs) are collected. PBSCs are collected beginning on day 10.

Patients receive high-dose melphalan IV on day -1. PBSCs are reinfused on day 0. G-CSF is administered IV or SC daily beginning on day 1 and continuing until blood counts recover. Between 8 and 14 weeks later, patients receive high-dose busulfan IV every 6 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2. PBSCs are reinfused on day 0 and G-CSF is administered IV or SC daily until blood counts recover.

Patients with responding or stable disease after chemotherapy receive maintenance therapy with interferon alfa beginning 14-20 weeks after day 0 of the second course of chemotherapy. Interferon alfa is administered SC 3 times a week for 3 years. Patients also receive pamidronate IV every 4 weeks until disease progression. Patients who are not in complete remission (CR) 6 months after completing the second course of chemotherapy receive oral thalidomide daily for a maximum of 1 year or for 3 months after achieving CR.

Patients are followed monthly for 1 year, every 3 months for 1 year, and then periodically thereafter.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study within approximately 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage I-III multiple myeloma

  * Less than 18 months since diagnosis
  * Smoldering myeloma allowed if there is evidence of progressive disease requiring therapy

    * At least 25% increase in M protein levels or Bence Jones excretion
    * Hemoglobin no greater than 10.5 g/dL
    * Hypercalcemia
    * Frequent infections
    * Rise in serum creatinine above normal on 2 separate occasions
  * Nonquantifiable monoclonal proteins allowed if other criteria for multiple myeloma or smoldering myeloma are met
* Response/status after induction therapy:

  * Responding or stable disease AND no greater than 40% myelomatous involvement of bone marrow
* No Waldenstrom's macroglobulinemia

PATIENT CHARACTERISTICS:

Age:

* 65 and under

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* Serum glutamic axaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) less than 2.5 times upper limit of normal
* Hepatitis B antigen or hepatitis C ribonucleaic acid (RNA) negative

Renal:

* See Disease Characteristics
* Creatinine no greater than 1.4 mg/dL
* Creatinine clearance greater than 65 mL/min

Cardiovascular:

* Cardiac ejection fraction at least 50% by multigated acquisition scan (MUGA) or echocardiogram

Pulmonary:

* Forced-expiratory volume in one second (FEV_1) greater than 60% of normal
* Diffusing capacity for carbon monoxide (DLCO) greater than 50% of predicted lower limit

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* Human immunodeficiency virus (HIV) negative
* No other medical or psychosocial problems that would increase patient risk
* No other malignancy within past 5 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix
* No known hypersensitivity to filgrastim (G-CSF) or Escherechi coli-derived proteins

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No more than 3 prior chemotherapy regimens
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 1999-04-13; Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Somlo, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Long-term Progression-free (PFS) and Overall Survival (OS) with Tandem Autologous Transplant (TASCT) After High-dose Induction With Melphalan (MEL) and Busulfan/cyclophosphamide (BU/CY), or a Novel Regimen of MEL and Total Marrow Irradiation (TMI), Followed by Maintenance With Interferon A-2 (IF) and/or Thalidomide (THAL). Haematologica 96(s1), 2011, s103. G. Somlo, J. Palmer, A. Dagis, M. O'Donnell, D. Snyder, F. Sahebi, N. Kogut, A. Brown, R. Spielberger, P.Parker, C. Karanes, L. Popplewell, A. Stein, A. Krishnan, J. Alvarnas, J. Wong, S. Forman.

RESULTS

PARTICIPANT FLOW:
Groups:
- High-dose Chemotherapy Followed by PBPC Rescue: Priming and Apheresis: Cyclophosphamide (CTX) 1.5 g/m2 and Filgrastim, 5 microgram/kg, t2x/day, until enough PBPC have been collected. This is day -10 to the first transplant.
  Cycle (transplant) 1: day -1: Melphalan 150 mg/m2 IV; day 0: reinfusion of half of the collected stem cells; day +1: Filgrastim 5 micrograms/kg/day IV until ANC>1000 per microliter.
  Day 0 of cycle 2 (C2) is at least 12 weeks and not past 18 weeks from day 1 of cycle 1. Day -8 C2: Start Dilantin 1000 mg IV. Days -7 through -4 of C2: Busulfan 0.8 mg/kg every 6 hours, 4 x per day. Dilantin 300 micrograms/day. Day -3 C2: CTX 60 mg/kg; start IV Mesna. Day -2 C2: CTX 60 mg/kg; continue Mesna IV. Day 0 C2: Reinfuse PBPC. Start Filgrastim 5 microgram/kg daily.
  12-18 weeks from day 0 of C2: alpha interferon 3 x 10 E 6 units/m2 3x per week (TIW) for 3 years.
  At 6 months following day 0 of C2, Thalidomide 400 mg/m2 will be administered orally to patients not in Complete Remission.
Period: Overall Study
Arm/Group | High-dose Chemotherapy Followed by PBPC Rescue
Started | 77
Completed | 68
Not Completed | 9
Not completed — No C2 given due to study on hold by IRB | 4
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- HD Chemo Followed by PBPC Rescue: HD Melphalan/Cyclophosphamide followed by PBPC Rescue, alpha-interferon, & pamidronate
Arm/Group | HD Chemo Followed by PBPC Rescue
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 75
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 54 [29 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 69
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 77
Stage of Multiple Myeloma [Count of Participants; unit: Participants] — Definitions are in section 4.0 "Staging Criteria" of the protocol: "Sequential High-Dose Melphalan and Busulfan/Cyclophosphamide Followed by Peripheral Blood Progenitor Cell Rescue, Interferon, Pamidronate, With or Without Thalidomide, for Patients with Multiple Myeloma"
  Stage I is Low Tumor Mass -- Indolent Myeloma Stage II is Intermediate Tumor Mass -- Smoldering Myeloma Stage III is High Tumor Mass
  Participants
    Stage I (Low Tumor Mass) | 6
    Stage II (Intermediate Tumor Mass) | 12
    Stage III (High Tumor Mass) | 50
    unrecorded | 9
M protein type [Count of Participants; unit: Participants]
  IgG | 36
  IgA | 22
  unrecorded | 19
Prior Anthracycline Chemotherapy [Count of Participants; unit: Participants]
  No | 6
  Yes | 62
  not recorded | 9

OUTCOME MEASURES:

1. Primary Outcome: Best Response Prior to Tandem Autologous Stem Cell Transplant
Description: Response gradations are specified in the "Blade criteria", Br J Haematol 1998; 102: 1115-1123. Serum myeloma protein is measured 2x at least six weeks apart, and urine M-component is measured 2x at least 3 weeks apart. Complete response (CR): less than 3% plasma cells in bone marrow or blood. Very good partial response (VGPR): Greater than 90% decrease in myeloma protein, and urine M-component less than 0.1 gm/day. Partial response (PR) Greater than 50% decrease in myeloma protein; urine M-component less than 0.2 gm/day. Lytic skeletal lesions must not increase, and serum calcium level must remain normal. Stable disease (SD): 25-49% decrease in protein and 25% decrease in urine M-component. Progressive disease (PD): Greater than 25% increase in myeloma protein, or hypercalcemia. Relapse: 1) increase greater than 100% of myeloma protein; 2) More than 25% increase of myeloma protein; 3) reappearance of the myeloma peaks; 4) increase in lytic bone lesions on radiographs.
Time Frame: From enrollment in the study until day -8: before dilantin given pre-first high-dose chemo preceeding first cycle of tandem autologous cell transplant
Measure: Count of Participants; unit: Participants
Groups:
- HD Chemo Followed by PBPC Rescue: Patients receive high-dose melphalan IV on day -1. PBSCs are reinfused on day 0. G-CSF is administered IV or SC daily beginning on day 1 and continuing until blood counts recover. Between 8 and 14 weeks later, patients receive high-dose busulfan IV every 6 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2. PBSCs are reinfused on day 0 and G-CSF is administered IV or SC daily until blood counts recover.
  filgrastim
  recombinant interferon alfa
  busulfan
  cyclophosphamide
  melphalan
  pamidronate disodium
  thalidomide
  peripheral blood stem cell transplantation
Arm/Group | HD Chemo Followed by PBPC Rescue
Number analyzed (Participants) | 68
Participants
  CR | 1
  VGPR | 4
  PR/SD | 62
  PD | 1

2. Primary Outcome: Response After Tandem Autologous Stem Cell Transplant
Description: as for outcome 1
Time Frame: After second cycle of tandem autologous stem cell transplant: Day 0 of second transplant to 12 weeks post-cycle 2 cell infusion of the tandem transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | HD Chemo Followed by PBPC Rescue
Number analyzed (Participants) | 65
Participants
  CR | 27
  VGPR | 11
  PR/SD | 24
  PD | 3

3. Primary Outcome: Three-year Overall Survival
Description: Kaplan-Meier estimate at three years post-first transplant of survival. Outcome is death or alive at follow-up (censored). 95 percent confidence interval of the point estimate is calculated using Greenwood's variance.
Time Frame: Estimate reported at three years after day 0 of the first cycle of infusion of cells of the tandem transplant.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | HD Chemo Followed by PBPC Rescue
Number analyzed (Participants) | 68
proportion of participants | 0.662 [0.536 to 0.761]

4. Primary Outcome: Progression-free Survival
Description: Kaplan-Meier estimate at three years post-first transplant of survival. Event of interest is the first of Death or Progression. Censoring is Alive in Continuous Complete Remission at date of last follow-up.
  95 percent confidence interval of the point estimate is calculated using Greenwood's variance.
Time Frame: Estimate reported at three years after day 0 of the first cycle of infusion of cells of the tandem transplant.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | HD Chemo Followed by PBPC Rescue
Number analyzed (Participants) | 68
proportion of participants | 0.456 [0.335 to 0.539]

5. Primary Outcome: Best Response at 6 Months Post Tandem Autologous Stem Cell Transplant
Description: as for outcome 1
Time Frame: Six months after day 0 of the first cycle of the tandem autologous stem cell transplant. This will be used to determine administration of thalidomide.
Measure: Count of Participants; unit: Participants
Arm/Group | HD Chemo Followed by PBPC Rescue
Number analyzed (Participants) | 63
Participants
  CR | 18
  VGPR | 5
  PR/SD | 29
  PD | 11

6. Primary Outcome: Best Response After Tandem Autologous Stem Cell Transplant and Maintenance
Description: as for outcome 1
Time Frame: Response after six months after day 0 of the first cycle of the tandem transplant, after administration of maintenance thalidomide if necessary, until three years post-day 0 of the first cycle of the tandem transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | HD Chemo Followed by PBPC Rescue
Number analyzed (Participants) | 16
Participants
  CR | 3
  VGPR | 1
  PR/SD | 6
  PD | 6

ADVERSE EVENTS:
Time Frame: From initial high dose (HD) chemotherapy up to three years post-initial HD chemotherapy, or death, or date taken off-study.
Description: When evaluating a toxicity, a modified National Cancer Institute (NCI) autologous bone marrow toxicity scale will be used.
Arm/Group | HD Chemo Followed by PBPC Rescue
All-Cause Mortality (participants affected / at risk) | 23/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 68/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HD Chemo Followed by PBPC Rescue (N=68)
Hemoglobin (Blood and lymphatic system disorders) | 7 (20)
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 7 (18)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3)
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 7 (30)
Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 7 (24)
Transfusion: Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 7 (11)
Transfusion: pRBCs for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 6 (9)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1 (2)
Palpitations (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (3)
Vasovagal episode (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 5 (7)
Hypotension (Cardiac disorders) | 2 (2)
Auditory/Ear - Other (Specify, __) AUDITORY/EAR CONGESTION (Ear and labyrinth disorders) | 1 (1)
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5)
Dehydration (Gastrointestinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Diarrhea associated with graft versus host disease (GVHD) (Gastrointestinal disorders) | 3 (5)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 4 (7)
Dysphagia, esophagitis, odynophagia (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 4 (5)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Specify, __) BENIGN PAPILLOMA (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Specify, __) DECREASED GASTRIC MOTILITY (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Specify, __) INCREASED SALIVA PRODUCTION (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Specify, __) TONGUE DISCOLORATION (Gastrointestinal disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 7 (17)
Proctitis (Gastrointestinal disorders) | 1 (1)
Salivary gland changes/saliva (Gastrointestinal disorders) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in the protocol. (Gastrointestinal disorders) | 7 (15)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3 (6)
Vomiting (Gastrointestinal disorders) | 7 (11)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 7 (19)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 6 (7)
Insomnia (General disorders) | 5 (8)
Rigors/chills (General disorders) | 2 (3)
Pain (General disorders) | 7 (35)
Pain - Other (Specify, __) ARM PAIN (General disorders) | 1 (1)
Pain - Other (Specify, __) BACK PAIN (General disorders) | 2 (2)
Pain - Other (Specify, __) BURNING SENSATION AROUND MOUTH (General disorders) | 1 (1)
Pain - Other (Specify, __) BURNING SENSATION IN MOUTH (General disorders) | 1 (1)
Pain - Other (Specify, __) JAW PAIN (General disorders) | 1 (1)
Pain - Other (Specify, __) LOW BACK PAIN (General disorders) | 1 (1)
Pain - Other (Specify, __) PAIN AT CATHETER SITE (General disorders) | 1 (1)
Pain - Other (Specify, __) SEVERE MOUTH PAIN (General disorders) | 1 (1)
Pain - Other (Specify, __) TOOTHACHE (General disorders) | 1 (1)
Hepatobiliary/Pancreas - Other (Specify, __) LOW ALKALINE PHOSPHATASE (Hepatobiliary disorders) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3 (4)
Graft versus host disease (Immune system disorders) | 1 (1)
Febrile neutropenia (fever without clinically or microbiologically documented infection) (Infections and infestations) | 1 (1)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 2 (4)
Infection, Viral (Infections and infestations) | 2 (2)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Weight gain - Veno-Occlusive Disease (VOD) for BMT studies if specified in the protocol. (Metabolism and nutrition disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 7 (19)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 7 (15)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 7 (16)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 7 (20)
Alkaline phosphatase (Metabolism and nutrition disorders) | 6 (13)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 7 (19)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 6 (12)
Creatinine (Metabolism and nutrition disorders) | 2 (4)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 7 (11)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3 (3)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 5 (7)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 7 (11)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 7 (12)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (6)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 3 (5)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (6)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 3 (4)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Mood alteration (Psychiatric disorders) | 6 (15)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatology/Skin - Other (Specify, __) DERMATOLOGY, SKIN OTHER (CHELIOSIS) (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other (Specify, __) DERMATOLOGY/ SI. ERYTHEMA AROUND HICKMAN (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 2 (2)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 (9)
Rash/desquamation associated with graft versus host disease (GVHD) (Skin and subcutaneous tissue disorders) | 6 (11)
Edema (Vascular disorders) | 5 (6)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Vascular disorders) | 1 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2004-02-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT00004088/Prot_SAP_000.pdf